CLINICAL TRIAL: NCT04617366
Title: Effect of Dynamic Individualized rTMS Based on fNIRS on Upper Limb Function of Stroke Patients
Brief Title: Dynamic Individualized rTMS Based on fNIRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJUFH-R-002
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Stroke; Rehabilitation; Repetitive Transcranial Magnetic Stimulation; Functional Near-infrared Spectroscopy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized rTMS strategy (Experimental): The individualized strategy will adjust the rTMS parameters promptly based on the results of fNIRS. This arm selects either the high-frequency rTMS to the contralesional dorsal premotor cortex (PMd) or the low-frequency rTMS to the contralesional primary motor cortex (M1) based on the lateralization index of the PMd measured by fNIRS.
  Interventions: Other: Individualized rTMS strategy
- Traditional rTMS strategy (Active Comparator): The control group will always be given low-frequency rTMS to contralesional M1.
  Interventions: Other: Traditional rTMS strategy

INTERVENTIONS:
Other: Individualized rTMS strategy — It will adjust the rTMS parameters based on the results of fNIRS.
  Arms: Individualized rTMS strategy
Other: Traditional rTMS strategy — The patients will always be given low-frequency rTMS to contralesional M1.
  Arms: Traditional rTMS strategy

SUMMARY:
Stroke patients do not respond well to the traditional repetitive transcranial magnetic stimulation (rTMS) strategy based on the competitive model. The studies found that the contralesional motion cortex has a compensatory effect on the realization of the motor function of the affected side-the compensatory model, and the degree of compensation will change as the function changes. The optimal neural regulation strategies under different models are opposite, so it is important to accurately evaluate which of the two models plays the leading role. And functional near-infrared spectroscopy (fNIRS) may accurately and quickly assess cortical function in order to determine the degree of participation of the contralesional motion cortex. We propose that the dynamic individualized strategy which adjust the rTMS parameters promptly based on the results of fNIRS will be better than the traditional stimulation strategy. This project will apply a blinded-assessment randomized controlled trial. The test group selects either the high-frequency rTMS to the contralesional dorsal premotor cortex (PMd) or the low-frequency rTMS to the contralesional primary motor cortex (M1) based on the lateralization index of the PMd measured by fNIRS. And the control group will always be given low-frequency rTMS to contralesional M1. The difference in the improvement of upper limb function between the two groups of patients was compared.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-79 years;
* Patients with first-onset subcortical infarcts within1 to 3 weeks after onset;
* TMS on the lesion side can induce motor evoked potential(MEP) of the abductor pollicis brevis muscle of the affected hand;
* Consciousness, sitting balance level 1 or above, can cooperate with assessment and treatment;
* The patient or its authorized agent signs the informed consent form.

Exclusion Criteria:

* Previous seizures;
* Suffered from mental illness such as depression, anxiety, mania, and schizophrenia before the stroke onset;
* Patients with metal on the head, cochlear implants, intracranial infections, etc. who are not suitable for rTMS.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer motor function score of upper limb | 3 months
  The score range is 0-66 points, the higher the score, the better the motor function of upper limb.

SECONDARY OUTCOMES:
Barthel index | 3 months
  The score range is 0-100 points, the higher the score, the better the activities of daily living.
Lateralization index (LI) | 3 months
  The LI score measured by fNIRS ranges from -1 to 1, with 1 indicating purely ipsilesional and -1 indicating purely contralesional activation.
Brain functional connection network | 3 months
  Using fNIRS to analyze the functional connection network between the motor areas of the bilateral cerebral hemispheres.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China